CLINICAL TRIAL: NCT05515081
Title: Two-Year Prospective Study of Antibody Response and Longevity Post SARS-CoV-2 Vaccine and Their Correlation With Humoral Factors
Brief Title: Antibody Response and Longevity Post SARS-CoV-2 Vaccine (SARS-AB)
Acronym: SARS-AB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021.06
Record Dates: First submitted 2022-08-18; First posted 2022-08-25 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2022-08

CONDITIONS: Vaccine Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- vaccinated healthy subject (Other): Procedure/Surgery: blood sample collection at regular intervals
  Interventions: Procedure: blood sample collection

INTERVENTIONS:
Procedure: blood sample collection — blood sample colletion at regular intervals

SUMMARY:
Longitudinal study on healthy subjects to investigate the longevity of the antibody response to the Pfizer-BioNTech COVID-19 vaccine. Venous blood samples will be collected on an outpatient basis from 400 adults at regular intervals (1, 2, 4, 6, 12, 18 and 24 months) after the second dose of the vaccine. In the event of the administration of a third dose, the participants already recruited will be subjected to a venous blood sample immediately before administration and subsequently at regular intervals (1, 2, 4, 6, 8 and 12 months). A laboratory serological test will be performed for each sample. The expression of humoral biomarkers will be evaluated with the Luminex methodology with the aim of identifying prognostic and predictive biomarkers of the response to the vaccine.

DETAILED DESCRIPTION:
Subject to informed consent, participants will be asked to provide a brief history of any previous SARS-CoV-2 infections and information on serological tests already performed. Subjects will undergo an outpatient venous blood sample at the San Camillo or Villa Salus hospital at regular intervals (1, 2, 4, 6, 12, 18 and 24 months) after the second dose of vaccine. Sample A will be pseudo-anonymized and the serological examination for the detection of antibodies will be carried out in the diagnostic laboratories of Villa Salus and / or in the Neurobiology laboratory of the San Camillo hospital. 5 cc of blood (sample B) will be taken separately and sent to the Neurobiology laboratory of the San Camillo hospital where they will be stored and analyzed in groups for the measurement of serum inflammation mediators (chemokines, cytokines) on a Luminex platform for analysis of a cytokine and chemokine panel (eg Cytokine & Chemokine Convenience 34-Plex Human ProcartaPlex ™ Panel 1). In the event that among the participants already recruited (200) there are individuals inoculated with a further dose of the vaccine, they will be subjected to a venous blood sample immediately before administration and subsequently at regular intervals (1, 2, 4, 6 , 8 and 12 months). The processing of the samples will take place in the manner described above.

ELIGIBILITY:
Inclusion Criteria:

• healthy adult subjects included in the vaccination program carried out for hospital staff of the San Camillo and Villa Salus hospitals in Venice starting from January 2021

Exclusion Criteria:

• none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-05-21 (Actual); Study Completion 2023-05-21 (Actual)

PRIMARY OUTCOMES:
Antibody titre assesssed by ELISA SARS-Cov-2 anti-RBD IgG kit | 12 months after 3rd dose
  Antibody levels at the same time points are compared by stratifying the sample into two groups based on whether or not volunteers had previously contracted the virus, using parametric (e.g., paired-sample t-test) or nonparametric (e.g., Wilcoxon test) tests depending on the distribution of the data.

SECONDARY OUTCOMES:
Cytokine measurement by ELISA test such as Cytokine & Chemokine Convenience 34-Plex Human ProcartaPlex ™ | 12 months after 3rd dose
  Correlation with humoral factors contributing to changes in the scale of the post-vaccination immune response will be performed with Pearson correlation test or Spearman correlation test as appropriated

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Camillo, Venice-Lido, Italy

IPD SHARING:
Plan to Share IPD: No